CLINICAL TRIAL: NCT00803452
Title: Lipids of the Human Tear Film and Their Effect on Tear Stability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Douglas Bourchman, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: lipidtearfilm; NEI RO-1- EY017094-02
Record Dates: First submitted 2008-12-01; First posted 2008-12-05 (Estimated); Results first posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Blepharitis
Keywords: Meibomian gland dysfunction; Lid margin disease; doxycycline; azithromycin; essential fatty acid
MeSH Terms: conditions — Blepharitis; Meibomian Gland Dysfunction | interventions — Doxycycline; Minocycline; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doxycycline (Active Comparator): Oral doxycycline
  Interventions: Drug: doxycycline
- azithromycin (Active Comparator): Topical azithromycin daily to the conjunctival culdesac
  Interventions: Drug: azithromycin

INTERVENTIONS:
Drug: doxycycline — Oral doxycycline 100mg bid
  Other Names: Minocycline
  Arms: Doxycycline
Drug: azithromycin — topical 1% azithromycin daily to eye
  Other Names: Azasite
  Arms: azithromycin

SUMMARY:
This prospective, randomized, comparative clinical trial evaluates the effect of either oral doxycycline, oral essential fatty acid, or topical azithromycin to modify the secretions of the meibomian gland in subjects with meibomian gland dysfunction and/or dry eye disease.

DETAILED DESCRIPTION:
Subjects with meibomian gland dysfunction undergo expression of the meibomian gland secretion prior to beginning treatment with either oral doxycycline or topical azithromycin solution. Doxycycline is dosed at 100 mg bid; topical azithromycin is delivered once per day as a 1% solution. Treatment with doxycycline is for two months; treatment with topical azithromycin is for one month. Following treatment, meibomian glands are again expressed and the lipids measured by spectroscopy (FTIR, MALDI-TOF, NMR)for characterization of structure and function. Analysis for presence of doxcycline or azithromycin is also performed. Changes in lipid parameters are correlated with clinical signs and symptoms of disease.

ELIGIBILITY:
Inclusion Criteria:

* Meibomian gland dysfunction

Exclusion Criteria:

* Lid margin scarring; herpetic blepharitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary N Foulks, MD, Principal Investigator — University of Louisville
Locations (1):
- Kentucky Lions Eye Center, Louisville, Kentucky, United States

REFERENCES:
- [Result] Foulks GN, Borchman D, Yappert M, Kakar S. Topical azithromycin and oral doxycycline therapy of meibomian gland dysfunction: a comparative clinical and spectroscopic pilot study. Cornea. 2013 Jan;32(1):44-53. doi: 10.1097/ICO.0b013e318254205f. PMID 22668581
- [Result] Foulks GN, Borchman D, Yappert M, Kim SH, McKay JW. Topical azithromycin therapy for meibomian gland dysfunction: clinical response and lipid alterations. Cornea. 2010 Jul;29(7):781-8. doi: 10.1097/ICO.0b013e3181cda38f. PMID 20489573
- [Derived] Borchman D, Foulks GN, Yappert MC, Bell J, Wells E, Neravetla S, Greenstone V. Human meibum lipid conformation and thermodynamic changes with meibomian-gland dysfunction. Invest Ophthalmol Vis Sci. 2011 Jun 1;52(6):3805-17. doi: 10.1167/iovs.10-6514. PMID 21398284

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Doxycycline | Azithromycin
Started | 9 | 22
Completed | 9 | 17
Not Completed | 0 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxycycline | Azithromycin | Total
Number analyzed (Participants) | 9 | 22 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (4) | 64 (3) | 65 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 10 | 10
  Male | 9 | 12 | 21
Region of Enrollment [Number; unit: participants]
  United States | 9 | 22 | 31

OUTCOME MEASURES:

1. Primary Outcome: Global Response to Therapy
Description: Global Response to Therapy (itch, dryness, burning and swelling of eyes) as assessed with a questionnaire completed by the subjects. The questionnaire asked subjects to rate their improvement on a scale from 4 to 0 with 4 being resolution of symptoms and 0 being no improvement. Data reported here represent the number of eye of subjects that reported that their symptoms were resolved or improved in each eye.
Time Frame: 4 weeks
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Doxycycline | Azithromycin
Number analyzed (Participants) | 9 | 22
Number analyzed (eyes) | 18 | 44
eyes | 16 | 41
Statistical Analysis 1: Comparison: Doxycycline vs Azithromycin; Test type: Superiority; p = .001, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Doxycycline | Azithromycin
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/22
Other Adverse Events (participants affected / at risk) | 0/9 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes